CLINICAL TRIAL: NCT01500083
Title: An Open-Label Expanded Access Trial for Bendamustine HCl in Patients With Indolent Non-Hodgkin's Lymphoma That Has Progressed During or Following Treatment With a Rituximab Regimen or Previously Untreated Chronic Lymphocytic Leukemia
Brief Title: Bendamustine Hydrochloride (HCl) in Indolent Non-Hodgkin's Lymphoma That Has Progressed During or Following Treatment With a Rituximab Regimen or Previously Untreated Chronic Lymphocytic Leukemia
Acronym: BENDACT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lundbeck Canada Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14293A
Record Dates: First submitted 2011-12-16; First posted 2011-12-26 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-06

CONDITIONS: Indolent Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia
Keywords: iNHL; CLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with Chronic Lymphocytic Leukemia (CLL) (Experimental): Patients with CLL will receive bendamustine at a dose of 100 mg/m2 on Days 1 and 2 in treatment cycles of 28 days for up to six cycles.
  Interventions: Drug: Bendamustine at a dose of 100 mg/m2
- Patients with Indolent Non-Hodgkin's Lymphoma (iNHL) (Experimental): Patients with iNHL will receive bendamustine at a dose of 120 mg/m2 on Days 1 and 2 in treatment cycles of 21 or 28 days for up to eight cycles.
  Interventions: Drug: Bendamustine at a dose of 120 mg/m2

INTERVENTIONS:
Drug: Bendamustine at a dose of 100 mg/m2 — Bendamustine will be administered intravenously over 30 minutes.
  Other Names: Treanda®
  Arms: Patients with Chronic Lymphocytic Leukemia (CLL)
Drug: Bendamustine at a dose of 120 mg/m2 — Bendamustine will be administered intravenous (i.v.) over 60 minutes.
  Other Names: Treanda®
  Arms: Patients with Indolent Non-Hodgkin's Lymphoma (iNHL)

SUMMARY:
The purpose of the current study is to evaluate additional safety data of bendamustine in up to 100 patients with Indolent Non-Hodgkin's Lymphoma (iNHL) relapsing from a rituximab regimen or Chronic Lymphocytic Leukemia (CLL). Patients will receive up to 6 or 8 cycles of bendamustine treatment using the dosing regimens of TREANDA® (bendamustine) approved in several countries, which have been shown to be reasonably well tolerated. The study protocol includes safety monitoring (i.e., adverse events, concomitant medications, supportive care, clinical safety laboratory tests, and clinical disease status monitoring).

It is an interventional, multicentre, prospective, open-label expanded access study, which in addition allows investigators in Canada, and their patients, access to bendamustine while it is pending Canadian marketing approval.

Although the treatment options available for patients with iNHL or CLL do induce substantial responses, there is no curative treatment. One potential drug candidate for the treatment of CLL and iNHL is bendamustine.

Bendamustine has been widely used in Germany for more than 30 years and is marketed in the United States for treatment of CLL and for treatment of iNHL that has progressed during or within 6 months of treatment with rituximab or a rituximab-containing regimen. In October 2010, the European Medicines Agency formally approved bendamustine in a number of Member States of the European Union for the treatment of patients with iNHL, CLL, and multiple myeloma. The drug's safety profile in these patient populations has been extensively characterized and no unexpected safety concerns are anticipated.

ELIGIBILITY:
Inclusion Criteria for iNHL:

* The patient has biopsy-confirmed diagnosis of indolent B-cell NHL documented as relapsed or refractory iNHL (following rituximab-based therapy).
* The patient has one of the following types of indolent B-cell lymphoma:

  * follicular lymphoma grade 1, 2, or 3A
  * marginal zone lymphoma
  * lymphoplasmacytic lymphoma
  * small lymphocytic lymphoma
* The patient has adequate haematologic function (unless abnormalities are related to lymphoma involvement of the bone marrow or hypersplenism caused by lymphoma).

Inclusion Criteria for CLL:

* The patient has previously confirmed (according to WHO criteria) untreated symptomatic chronic B-cell lymphocytic leukemia Binet Stage B or Binet Stage C or Rai stage II to IV in need of medical treatment.
* The patient has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.

Exclusion Criteria:

* The patient has participated in a clinical study <30 days prior to the Screening Visit.
* The patient has one or more of the following conditions:

  * active transformed lymphoma
  * any history of central nervous system or leptomeningeal lymphoma
  * an active malignancy other than the target cancer within the past 5 years
  * human immunodeficiency virus
* The patient is, in the investigator's opinion, unlikely to comply with the protocol or is unsuitable for any reason.

Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (16):
- Canada (16):
  - CA015, Calgary, Alberta
  - CA014, Edmonton, Alberta
  - CA016, Kelowna, British Columbia
  - CA011, Vancouver, British Columbia
  - CA013, Victoria, British Columbia
  - CA012, Winnipeg, Manitoba
  - CA004, Halifax, Nova Scotia
  - CA009, Brampton, Ontario
  - CA003, Hamilton, Ontario
  - CA002, Ottawa, Ontario
  - CA006, Toronto, Ontario
  - CA005, Windsor, Ontario
  - CA001, Montreal, Quebec
  - CA010, Montreal, Quebec
  - CA007, Saskatoon, Saskatchewan
  - CA008, Québec

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Previously Untreated CLL: Patients with CLL will receive bendamustine at a dose of 100 mg/m2 on Days 1 and 2 in treatment cycles of 28 days for up to six cycles. Bendamustine will be administered i.v. over 30 minutes.
- Patients With iNHL: Patients with iNHL will receive bendamustine at a dose of 120 mg/m2 on Days 1 and 2 in treatment cycles of 21 or 28 days for up to eight cycles. Bendamustine will be administered intravenous (i.v.) over 60 minutes.
Period: Overall Study
Arm/Group | Patients With Previously Untreated CLL | Patients With iNHL
Started | 16 | 74
Completed | 4 | 31
Not Completed | 12 | 43
Not completed — Adverse Event | 4 | 17
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal of Consent | 0 | 1
Not completed — Disease Progression | 2 | 10
Not completed — Investigator Discretion | 3 | 8
Not completed — Other Reasons | 2 | 5

BASELINE CHARACTERISTICS:
Population: all-patients-treated set (APTS): all enrolled patients who took at least one dose of investigational medicinal product (IMP)
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Previously Untreated CLL | Patients With iNHL | Total
Number analyzed (Participants) | 16 | 74 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (7.12) | 63.1 (10.84) | 64.2 (10.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 35 | 44
  Male | 7 | 39 | 46

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events
Time Frame: Up to 266 days
Population: APTS
Measure: Number; unit: number of adverse events
Arm/Group | Patients With Previously Untreated CLL | Patients With iNHL
Number analyzed (Participants) | 16 | 74
number of adverse events | 298 | 302

ADVERSE EVENTS:
Time Frame: Up to 266 days
Arm/Group | Patients With Previously Untreated CLL | Patients With iNHL
Serious Adverse Events (participants affected / at risk) | 6/16 | 27/74
Other Adverse Events (participants affected / at risk) | 16/16 | 72/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Previously Untreated CLL (N=16) | Patients With iNHL (N=74)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 3 | 6
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Bronchopneumonia (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Nocardiosis (Infections and infestations) | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 2
Pneumonia (Infections and infestations) | 0 | 3
Toxic shock syndrome (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 1 | 2
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Previously Untreated CLL (N=16) | Patients With iNHL (N=74)
Anaemia (Blood and lymphatic system disorders) | 4 | 17
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2
Haemolysis (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 3
Neutropenia (Blood and lymphatic system disorders) | 5 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 14
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2
Tachycardia (Cardiac disorders) | 1 | 2
Vertigo (Ear and labyrinth disorders) | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 2 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 3
Anal pruritus (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 5 | 23
Diarrhoea (Gastrointestinal disorders) | 9 | 21
Dry mouth (Gastrointestinal disorders) | 2 | 10
Dyspepsia (Gastrointestinal disorders) | 1 | 15
Dysphagia (Gastrointestinal disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 4
Mouth ulceration (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 12 | 50
Reflux gastritis (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 7
Vomiting (Gastrointestinal disorders) | 9 | 26
Asthenia (General disorders) | 2 | 5
Chest pain (General disorders) | 2 | 4
Chills (General disorders) | 3 | 11
Fatigue (General disorders) | 8 | 43
Infusion related reaction (General disorders) | 1 | 3
Injection site phlebitis (General disorders) | 1 | 0
Malaise (General disorders) | 2 | 2
Mucosal inflammation (General disorders) | 0 | 4
Oedema peripheral (General disorders) | 2 | 12
Pain (General disorders) | 1 | 2
Pyrexia (General disorders) | 4 | 21
Cystitis (Infections and infestations) | 1 | 0
Eye infection (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 6
Nasopharyngitis (Infections and infestations) | 2 | 1
Rhinitis (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Skin infection (Infections and infestations) | 1 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 5
Urinary tract infection (Infections and infestations) | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 2
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 2 | 1
Blood magnesium decreased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 1
Gamma-glutamyltransferase increased (Investigations) | 2 | 1
Haemoglobin decreased (Investigations) | 0 | 6
Haptoglobin decreased (Investigations) | 1 | 0
Lymphocyte count decreased (Investigations) | 2 | 1
Neutrophil count decreased (Investigations) | 4 | 7
Platelet count decreased (Investigations) | 2 | 11
Weight decreased (Investigations) | 2 | 9
White blood cell count decreased (Investigations) | 2 | 6
Decreased appetite (Metabolism and nutrition disorders) | 4 | 20
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperchloraemia (Metabolism and nutrition disorders) | 3 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 6
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 7
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 6
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 4
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ageusia (Nervous system disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 2
Disturbance in attention (Nervous system disorders) | 1 | 3
Dizziness (Nervous system disorders) | 2 | 13
Dysgeusia (Nervous system disorders) | 0 | 17
Headache (Nervous system disorders) | 5 | 17
Anxiety (Psychiatric disorders) | 2 | 4
Insomnia (Psychiatric disorders) | 0 | 6
Dysuria (Renal and urinary disorders) | 1 | 1
Micturition urgency (Renal and urinary disorders) | 1 | 1
Pollakiuria (Renal and urinary disorders) | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 13
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 8
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 2
Erythema (Skin and subcutaneous tissue disorders) | 1 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 7
Rash (Skin and subcutaneous tissue disorders) | 2 | 8
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 1
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0
Hot flush (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypotension (Vascular disorders) | 1 | 4
Phlebitis (Vascular disorders) | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of this study will be published. Authors of the primary publication based on this study must fulfil the criteria defined by the International Committee of Medical Journal Editors (ICMJE). The primary publication must be published before any secondary publications are submitted for publication.